CLINICAL TRIAL: NCT06981156
Title: Evaluation of the Neurologic Assessment in Pediatric Neuro-Oncology (pNANO)
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0533; A536755 (Other: UW Madison); Protocol Version 3/14/25 (Other: UW Madison); UW24162 (Registry Identifier: OnCore ID); NCI-2025-03504 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Brain Tumor; Pediatric Spine Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Brain and Spine Tumor Patients
  Interventions: Diagnostic Test: pNANO Assessment

INTERVENTIONS:
Diagnostic Test: pNANO Assessment — pNANO assesses patient gait, strength, cerebellar function, visual fields, visual acuity, facial strength, level of consciousness, extraocular movement, dysarthria, and dysphagia
  The patient will be assessed by 2-3 different clinicians during each of 2 visits.
  Other Names: Pediatric Neuro-Oncology

SUMMARY:
This study aims to investigate a neurologic exam scale to provide an objective and more standard way to assess tumor response in pediatric patients with brain and spinal cord tumors.

DETAILED DESCRIPTION:
This study is designed to evaluate inter-observer variability of the pNANO scale when implemented during routine clinic visits for pediatric brain and spine tumor patients. Typically, during a routine clinic visit for patients with pediatric brain and spine tumors, a neurological examination is completed and documented by a provider in clinic notes under the section 'Physical examination', sub-heading 'Neurologic examination.'

For this study, every participant will have neurologic examinations performed by 2 or 3 (if feasible), separate providers on the same day (patient's scheduled provider and one or two additional providers from the Study Team), during a scheduled, routine clinic visit(s). To allow for potential significant discrepancies in exams between two providers, if feasible, a third provider will complete an examination at each visit. Each provider will independently perform the neurologic examination and will document the findings on the pNANO scale scorecard.

Each provider will also record the amount of time it took to complete their neurologic examination. The providers will not communicate with each other about the findings and will be completely blinded to each other's evaluations.

The pNANO scale will be completed at a second clinic visit, between 1-6 months out from the initial assessment. Telemedicine visit evaluations will be allowed for 20% of patients enrolled on study to assess if this scale is feasible via telemedicine. For telemedicine visits, one provider will need to be in clinic to complete the first examination and the second provider will be virtual to complete the second examination on the same day. A third provider would need to be in clinic to complete an examination.

For the second evaluation 1-6 months after the first, the same will apply, one or two providers in clinic to complete the first examination while the second/third provider will be virtual. Providers can include physicians and advanced practice providers of any subspecialty: neurology, hematology-oncology, radiation oncology, neurosurgery, physical medicine and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 1 year old
* must be seen in the pediatric clinic
* Radiographic or histologic confirmation of a brain or spine tumor at the time of initial diagnosis
* Patient or parent/guardian must be able to understand the consent and be willing to sign a written informed consent document according to institutional guidelines.

Exclusion Criteria:

* none specified

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric brain or spine tumor patients greater than or equal to 1 year old.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Inter-observer Variability in pNANO Scores: Difference in Mean Cumulative Scores | Visit 1 (baseline), Visit 2 (up to 6 months)
  The Pediatric Neurologic Assessment in Neuro-Oncology (pNANO) is scored in multiple domains: - strength, level of consciousness, and gait domains (each individually scored 0-3)
  * facial strength, cerebellar function, visual fields, extraocular movements, dysphagia, and dysarthria domains (each individually scored 0-2)
  * visual acuity domain scored from 0-1 If summed, cumulative scores range from 0 (normal) to 22 (inability to function in each relevant domain)
  Investigators will explore variability across all domains.

SECONDARY OUTCOMES:
Feasibility: Clinical Exams that may correlate with pNANO scores | Visit 1 (baseline), Visit 2 (up to 6 months)
  Investigators will explore whether pNANO scores (individual domains or cumulative scores) correlate with clinical exams.
Feasibility: Inter-observer variability of pNANO scores between in clinic visits and Telemedicine reported as Difference in Mean Cumulative Scores | Visit 1 (baseline), Visit 2 (up to 6 months)
  A subset of participants (approximately 20%) will be assessed remotely to study any impact telemedicine has on pNANO scoring. If summed, cumulative scores range from 0 (normal) to 22 (inability to function in each relevant domain).
  Investigators will explore variability across all domains.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Stuckert, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- American Family Children's Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No